CLINICAL TRIAL: NCT00846027
Title: An Open Label Study to Assess the Effect of First Line Treatment With Avastin in Combination With Paclitaxel and Gemcitabine in Progression-free Survival in Patients With HER-2 Negative Breast Cancer
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Taxane-based Chemotherapy as First Line Treatment in Patients With HER-2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21999; 2008-003657-32 (EudraCT Number)
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel; Gemcitabine

ARMS (1):
- Bevacizumab + paclitaxel + gemcitabine (Experimental): Participants received bevacizumab 10 mg/kg intravenously (IV), paclitaxel 150 mg/m^2 IV, and gemcitabine 2000 mg/m^2 IV on Day 1 and Day 15 of each 4-week cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was supplied as a sterile liquid in glass vials.
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel was supplied as a sterile liquid in glass vials.
  Other Names: Taxol
Drug: Gemcitabine — Gemcitabine was supplied as a sterile liquid in glass vials.
  Other Names: Gemzar

SUMMARY:
This single-arm study assessed the efficacy and safety of first-line treatment with Avastin (bevacizumab) in combination with taxane-based chemotherapy (paclitaxel and gemcitabine) in patients with HER-2 negative breast cancer. Patients received Avastin 10 mg/kg iv, paclitaxel 150 mg/m^2 iv, and gemcitabine 200 mg/m^2 iv on Day 1 and Day 15 of each 4-week treatment cycle until disease progression, death, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, ≥ 18 years of age.
* Breast cancer, with measurable, locally recurrent or metastatic lesions, or patients with bone metastasis only.
* HER-2 negative disease.
* Candidates for chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.

Exclusion Criteria:

* Previous chemotherapy for metastatic or locally advanced breast cancer.
* Previous radiotherapy for treatment of metastatic breast cancer.
* Any prior adjuvant treatment with anthracyclines completed < 6 months prior to enrollment.
* Chronic daily treatment with corticosteroids (≥ 10 mg/day), aspirin (> 325 mg/day) or clopidogrel (> 75mg/day).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Spain (19):
  - Elda, Alicante
  - Barcelona, Barcelona
  - Manresa, Barcelona
  - Burgos, Burgos
  - Cadiz, Cadiz
  - Córdoba, Cordoba
  - Granada, Granada
  - Huelva, Huelva
  - Jaén, Jaen
  - Las Palmas de Gran Canaria, Las Palmas
  - Lugo, Lugo
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Marbella, Malaga
  - Murcia, Murcia
  - Vigo, Pontevedra
  - Seville, Sevilla
  - Sagunto, Valencia
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab + Paclitaxel + Gemcitabine
Started | 90
Received Treatment | 83
Completed | 0
Not Completed | 90
Not completed — Death | 3
Not completed — Disease Progression | 30
Not completed — Toxicity | 12
Not completed — Patient Decision | 7
Not completed — Investigator Discretion | 29
Not completed — Protocol Violation | 2
Not completed — Subject Not Treated | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All participants enrolled in the study.
Arm/Group | Bevacizumab + Paclitaxel + Gemcitabine
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.20 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from enrollment in the study to the first documented disease progression using Response Evaluation Criteria In Solid Tumors (RECIST) or death from any cause, whichever occurred first.
Time Frame: Baseline to the end of the study (up to 2 years 10 months)
Population: Intent-to-treat population: All participants who were enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Paclitaxel + Gemcitabine
Number analyzed (Participants) | 90
Months | 11.51 [9.01 to 17.59]

2. Secondary Outcome: Percentage of Participants With an Objective Response
Description: An objective response was defined as a complete or partial response determined on 2 consecutive occasions ≥ 4 weeks apart using Response Evaluation Criteria in Solid Tumors (RECIST). Complete response was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must be < 10 mm on the short axis. Partial response was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum.
Time Frame: Baseline to the end of the study (up to 2 years 10 months)
Population: Intent-to-treat population: All participants who were enrolled in the study. Only participants who had a response evaluation were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab + Paclitaxel + Gemcitabine
Number analyzed (Participants) | 76
Percentage of participants | 72.37 [60.91 to 82.01]

3. Secondary Outcome: Duration of the Objective Response
Description: Duration of the objective response is defined as the time from a complete or partial response to disease progression or death due to disease.
Time Frame: Baseline to the end of the study (up to 2 years 10 months)
Population: Intent-to-treat population: All participants who were enrolled in the study. Only participants who had a response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Paclitaxel + Gemcitabine
Number analyzed (Participants) | 55
Months | 12.39 [7.63 to 15.16]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the first dose of study medication until death.
Time Frame: Baseline to the end of the study (up to 2 years 10 months)
Population: Intent-to-treat population: All participants who were enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Paclitaxel + Gemcitabine
Number analyzed (Participants) | 90
Months | 27.39 [21.86 to NA] — The upper limit of the confidence interval could not be calculated due to too few events.

ADVERSE EVENTS:
Description: Safety population: All enrolled participants who receive at least 1 dose of medication and who satisfied all inclusion criteria and none of the exclusion criteria. 7 participants did not receive at least 1 dose of medication and 1 participant did not satisfy an inclusion criterion. These 8 participants were not included in the safety population.
Arm/Group | Bevacizumab + Paclitaxel + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 21/82
Other Adverse Events (participants affected / at risk) | 82/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel + Gemcitabine (N=82)
Anorexia (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Fever (Infections and infestations) | 4
Catheter site infection (Infections and infestations) | 2
Febrile neutropenia (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1
Neutrophils count decreased (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel + Gemcitabine (N=82)
Nausea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 20
Constipation (Gastrointestinal disorders) | 13
Anorexia (Gastrointestinal disorders) | 10
Dysgeusia (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 4
Distension/bloating, abdominal (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Periodontal disease (Gastrointestinal disorders) | 2
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Perforation, GI (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Dental: teeth (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Pain oral-gums (General disorders) | 28
Pain muscle (Musculoskeletal and connective tissue disorders) | 18
Pain abdomen (Gastrointestinal disorders) | 13
Pain joint (Musculoskeletal and connective tissue disorders) | 12
Pain back (Musculoskeletal and connective tissue disorders) | 9
Pain head/headache (Nervous system disorders) | 7
Pain extremity limb (General disorders) | 5
Pain bladder (Renal and urinary disorders) | 3
Pain, other (General disorders) | 3
Pain bone (Musculoskeletal and connective tissue disorders) | 3
Chest/thorax (General disorders) | 2
Pain other back (Musculoskeletal and connective tissue disorders) | 1
Pain abdomen (Gastrointestinal disorders) | 1
Pain neck (Musculoskeletal and connective tissue disorders) | 1
Pain uterus (Gastrointestinal disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 28
Rash/desquamation (Skin and subcutaneous tissue disorders) | 20
Nail changes (Skin and subcutaneous tissue disorders) | 17
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 7
Dermatology/skin, other (Skin and subcutaneous tissue disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 4
Hand-foot (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 1
Alteration in scarring (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 54
Fever (General disorders) | 15
Hot flashes (Vascular disorders) | 1
Constitutional symptoms, other (General disorders) | 2
Insomnia (Psychiatric disorders) | 1
Diaphoresis (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 62
Mood alteration (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 4
Confusion (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Neuropathy: cranial optic (Nervous system disorders) | 1
Neutrophils low (Blood and lymphatic system disorders) | 26
Haemoglobin decreased (Blood and lymphatic system disorders) | 15
Platelets low (Blood and lymphatic system disorders) | 6
Leukocytes low (Blood and lymphatic system disorders) | 6
Blood/bone marrow , other (Blood and lymphatic system disorders) | 3
Haemorrhage, pulmonary/upper respiratory nose (Vascular disorders) | 30
Haemorrhage, gastrointestinal oral cavity (Vascular disorders) | 4
Haemorrhage, gastrointestinal rectum (Vascular disorders) | 2
Haemorrhage, genitourinary bladder (Vascular disorders) | 2
Haemorrhage, pulmonary/upper respiratory lung (Vascular disorders) | 2
Haemorrhage/bleeding, other (Vascular disorders) | 1
Haemorrhage, gastrointestinal varices (rectal) (Vascular disorders) | 1
Haemorrhage, genitourinary uterus (Vascular disorders) | 1
Infection bladder (urinary) (Infections and infestations) | 5
Infection - other nose (Infections and infestations) | 4
Infection with unknown absolute neutrophil count (Infections and infestations) | 4
Infection, other (Infections and infestations) | 4
Infection - other general catheter-related (Infections and infestations) | 3
Infection other conjunctiva (Infections and infestations) | 3
Infection pharynx (Infections and infestations) | 3
Febrile neutropenia (Infections and infestations) | 2
Infection - other general oral cavity-gums (Infections and infestations) | 2
Infection sexual/reproductive function vaginal (Infections and infestations) | 1
Infection vaginal (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Dysarthria (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Nasal/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Cardiac disorders) | 13
Left ventricular systolic dysfunction (Cardiac disorders) | 2
Cardiac ischemia/infarction (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Pulmonary hypertension (Cardiac disorders) | 1
Proteinuria (Investigations) | 3
Alanine transaminase, serum glutamic pyruvic transaminase (Investigations) | 2
Aspartate aminotransferase (Investigations) | 2
Metabolic, other (Investigations) | 2
Alanine transaminase/aspartate aminotransferase high (Investigations) | 1
Uric acid, serum-high (Investigations) | 1
Alanine transaminase (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
Oedema: limb (Metabolism and nutrition disorders) | 8
Lymphatics - other lymphangitis (Metabolism and nutrition disorders) | 1
Watery eye (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Ocular/visual (Eye disorders) | 1
Ophthalmoplegia/diplopia (Eye disorders) | 1
Irregular menses (Endocrine disorders) | 2
Sexual/reproductive, other (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Cystitis (Renal and urinary disorders) | 2
Bladder spasms (Renal and urinary disorders) | 1
Allergic reaction/hypersensitivity (Immune system disorders) | 2
Allergic reaction (Immune system disorders) | 1
Muscle weakness- extremity lower (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1
Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 1
Secondary malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hot flashes (Endocrine disorders) | 1
Phlebitis (Vascular disorders) | 1
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.